CLINICAL TRIAL: NCT02580994
Title: REACTION: A Phase II Study of Etoposide and Cis/Carboplatin With or Without Pembrolizumab in Untreated Extensive Small Cell Lung Cancer
Brief Title: Pembrolizumab in Untreated Extensive SCLC
Acronym: REACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1417-LCG; 2014-003090-42 (EudraCT Number)
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Extended Disease Small Cell Lung Cancer; phase II; randomized; pembrolizumab; cross-over; etoposide; cisplatin; carboplatin; rechallenge
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pembrolizumab; Etoposide; Cisplatin; Carboplatin; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + chemotherapy (Experimental): Pembrolizumab, in combination with cis/carboplatin and etoposide for 4 cycles intravenous 200mg on day 1 (every 3 weeks), pembrolizumab continued alone as continuation maintenance until progressive disease
  Interventions: Drug: Pembrolizumab; Drug: cis/carboplatin and etoposide
- Chemotherapy (Active Comparator): 4 cycles of cis/carboplatin and etoposide
  Interventions: Drug: cis/carboplatin and etoposide

INTERVENTIONS:
Drug: Pembrolizumab — IV infusion at the dose of 200 mg on day 1 every 3 weeks
  Other Names: MK-3475; Keytruda
  Arms: Pembrolizumab + chemotherapy
Drug: cis/carboplatin and etoposide — Cisplatin 80 mg/m2 or Carboplatin Area Under the Curve (AUC) 5 IV infusion on day 1 Etoposide 100 mg/m2 IV infusion on day 1, 2 and 3
  Other Names: Platinol, Paraplatin and Etopophos

SUMMARY:
This is a multicenter, open-label, two armed, controlled, and randomized phase II trial investigating the activity of pembrolizumab in combination with standard chemotherapy in Extensive Disease (ED)-SCLC.

DETAILED DESCRIPTION:
This is a multicenter, open-label, two armed, controlled, and randomized phase II trial investigating the activity of pembrolizumab in combination with standard chemotherapy in ED-SCLC.

Extended stage Small Cell Lung Cancer (SCLC) patients will be registered, after signing the informed consent, and then centrally randomized 1:1 to the experimental arm (Arm A) and the control arm (Arm B).

Cross-over at the time of disease progression will be allowed for arm B only.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC
* Extended disease according to the criteria of the Veteran's Administration - Lung Cancer Group (VALG): disease extended beyond a hemithorax and the supraclavicular node area. Pleural involvement will be considered as extended disease
* Assessment of adequate tissue availability for Program Cell Death-Ligand 1 (PD-L1) immunohistochemistry testing
* Before patient registration, written informed consent must be given according to International Conference of Harmonization-Good Clinical Practice (ICH-GCP), and national/local regulations
* Tumor assessment performed within 10 days before randomization. Patient may or may not have measurable disease
* Previous palliative brain radiotherapy is allowed if terminated at least 3 weeks before randomization
* Partial or complete response according to RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 after 2 cycles of any platinum-based induction chemotherapy regimen
* Adequate hematopoietic, hepatic and renal function within 10 days before randomization defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10E9/L, Hemoglobin (Hb) ≥ 9 g/dL and platelet count ≥ 100 x 10E9/L
  * Serum creatinine clearance ≥ 60 mL/min as calculated with Cockcroft-Gault formula
  * Bilirubin ≤ 1.5 x Upper Limit Normal (ULN), Alanine Aminotransferase (ALT) (SGTP) and Aspartate Transaminase (AST) (SGOT) ≤ 3 x ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as a PTT is within therapeutic range of intended use of anticoagulants N.B. Lactate Dehydrogenase (LDH) level assessment is mandatory for randomization
* Women of child bearing potential (WOCBP) must have a negative urine or serum pregnancy test within 72 hours before randomization
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by investigator, during the study treatment period and for at least 120 days after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing before randomization and until 120 days after the last study treatment

Exclusion Criteria:

* Prior systemic therapy for SCLC; previous treatment with platinum and etoposide concomitant with radiotherapy (RT) for limited disease is allowed if terminated at least 1 year before patient randomization
* known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (i.e. without evidence of progression by imaging and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not received steroids for at least 7 days before randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 3-4 (at registration) (patients who are judged by the investigator to be PS 2 due to primary disease are the only PS 2 patients who are eligible)
* ECOG PS 2-4 (at randomization)
* Less than 3 month life expectancy
* History of interstitial lung disease (ILD) or a history of (non-infectious) pneumonitis that required oral or IV steroids (other than Chronic Obstructive Pulmonary Disease [COPD] exacerbation) or current pneumonitis or current evidence of ILD
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs), any replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Previous allogeneic tissue/solid organ transplant
* Active infection requiring therapy
* Known history of Human Immunodeficiency Virus (HIV) (known HIV 1/2 antibodies positive). No known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg results. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative Hepatitis C Virus (HCV) RNA results greater than the lower limits of detection of the assay
* Ongoing grade ≥ 2 peripheral neuropathy
* Prior treatment with platinum, anti-PD-1, anti-PD-L1/2, anti interleukin-7 receptor-alpha (anti-CD127), Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4) modulators
* Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the 3 days before randomization:
* Corticosteroid use on study for management of pembrolizumab Events of Clinical Interest (ECIs), as pre-medication for the administration of chemotherapies, and/or a pre-medication for contrast allergies/reactions is allowed
* Daily prednisone at doses of 5-7.5 mg is allowed as an example of replacement therapy. Equivalent hydrocortisone doses are also permitted if administered as a replacement therapy
* Prior use of live vaccines within 30 days before randomization. Examples of live vaccines include, but are not limited to, the following : measles, mumps, rubella, chicken pox, shingles, yellow fever, influenza A virus subtype (H1N1) flu, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine
* Presence of any clinical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Concurrent treatment with any investigational agent within 4 weeks before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Increase in Progression Free Survival | 6 months

SECONDARY OUTCOMES:
Overall Survival | 12 months

CONTACTS AND LOCATIONS:
Locations (18):
- France (10):
  - Centre Hospitalier d'Avignon - Hopital Duffaut, Avignon
  - CHU de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Hopitalier Intercommunal De Creteil, Créteil
  - Centre Leon Berard, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hopital Nord, Marseille
  - Centre Hospitalier D'Annecy, Metz-Tessy
  - Assistance Publique - Hopitaux de Paris - Hopital Avicenne, Paris
  - Centre Paul Strauss, Strasbourg
  - Gustave Roussy, Villejuif
- Italy (6):
  - Ospedale Cannizzaro, Catania
  - Santa Croce e Carle General Hospital, Cuneo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Paolo, Milan
  - Ospedale S. Luigi Gonzaga - Universita Di Torino, Orbassano
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield